CLINICAL TRIAL: NCT06485193
Title: Det medfødte Immunforsvar og Det Enteriske Nervesystem Ved Crohns Sygdom
Brief Title: The Innate Immune Response and Enteric Nervous System in Crohn's Disease.
Status: Terminated | Type: Observational
Why Stopped: Preliminary results showed no signs of associations in the data.
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Thomsen, MD, Aalborg University Hospital
Other Study IDs: N-20230024
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Immunohistochemical analysis of archived diagnostic tissue samples.

SUMMARY:
The study aims to explore the relationships between inflammation, nerve changes, and the expression of interferon-stimulated proteins in inflamed and non-inflamed bowel areas from patients with Crohn's disease. Crohn's disease is a chronic inflammatory condition with complex causes and mechanisms that remain uncertain despite extensive research.

Methods and Procedures This exploratory study utilizes tissue samples from a clinical biobank at Aalborg University Hospital. The samples are paraffin-embedded blocks from which tissue sections are prepared for immunohistochemical and histological staining. The study focuses on assessing the expression of interferon-stimulated proteins through optimized immunohistochemical staining methods, ensuring reproducibility via automated machines. The protein expressions are then analyzed qualitatively and semi-quantitatively and compared with structural changes in the bowel tissues.

ELIGIBILITY:
Inclusion Criteria:

* Histological preparations (tissue samples) from patients with Crohn's disease who have undergone bowel resection at Aalborg University Hospital in the period from 2012 to 2023.

Exclusion Criteria:

* If the tissue material does not include the ileocecal region.
* If the pathology report does not indicate that there is tissue material from both inflamed and non-inflamed areas.
* If the patient has registered a prohibition against research in the Tissue Utilization Registry.
* The selection of cases starts with the most recent (by date) and stops when 25 suitable cases are found.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
MxA expression | June 1 2024
  Immunohistochemical Mxa expression

SECONDARY OUTCOMES:
Enterovirus positivity | June 1 2024
  pan-enterovirus immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Northern Region, Denmark

IPD SHARING:
Plan to Share IPD: No